CLINICAL TRIAL: NCT07044830
Title: Obstructive Sleep Apnea Treatment From Acute to Chronic Phase of Stroke - A Randomized Clinical Trial
Brief Title: Obstructive Sleep Apnea Treatment From Acute to Chronic Phase of Stroke
Acronym: ATACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital das Clínicas de Ribeirão Preto (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); ResMed Foundation (Other)
Responsible Party: Principal Investigator, Millene Rodrigues Camilo, Principal Investigator, Hospital das Clínicas de Ribeirão Preto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20802619.2.0000.5440
Record Dates: First submitted 2025-06-01; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke; Obstructive Sleep Apnea
Keywords: Stroke; Obstructive Sleep Apnea; Sleep
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea, Obstructive; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Severe OSA treated (Active Comparator): AHI≥30: treated with CPAP
  Interventions: Device: CPAP
- Severe OSA untreated (No Intervention): AHI≥30: without CPAP
- No OSA (No Intervention): AHI<5
- Mild OSA (No Intervention): 5≥AHI<15
- Moderate OSA (No Intervention): 15≤AHI<30

INTERVENTIONS:
Device: CPAP — Automatically-adjusting continuous positive airway pressure (CPAP)
  Arms: Severe OSA treated

SUMMARY:
The study aims to evaluate whether early treatment of obstructive sleep apnea with continuous positive airway pressure in ischemic stroke patients has a favorable effect on functional recovery.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is present in more than 70% of acute stroke patients, and has been related to poor short-and long-term outcomes. The treatment of choice for OSA is continuous positive airway pressure (CPAP).

The objective of this prospective, multicenter, randomized study is to evaluate the impact of CPAP treatment on clinical outcomes in post-stroke patients. Respiratory polygraphy will be performed in all eligible participants, and those with severe OSA will be randomized to receive either CPAP therapy or conservative management. CPAP use will initiated within the first 48-72 hours of hospital admission and continued through 2 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial non-lacunar ischemic stroke, including anterior, middle, and posterior cerebral artery territories
* Aged 18 to 80 years
* Symptom onset or symptom recognition to admission < 12 hours
* NIHSS score ≥ 4 and ≤ 20 at enrollment
* Signed informed consent form obtained from the participant or their legal representative

Exclusion Criteria:

* Prior stroke
* Previous diagnosis of OSA with current CPAP use or previously failed CPAP
* Pre-stroke disability (mRS > 1)
* Coma or stupor
* Orotracheal intubation
* Clinical instability or severe pre-existing illness (e.g., heart failure, oxygen-dependent COPD, renal or hepatic failure)
* Psychomotor agitation
* High likelihood of neurosurgical intervention within the first 48 hours
* Oxygen therapy >2 L/min
* Known severe neurological disease (e.g., dementia, Parkinson's disease, multiple sclerosis, or other neurodegenerative conditions)
* Chronic alcohol or drug use with high risk of withdrawal during hospitalization
* Pregnant or suspected pregnant women
* Inability to complete follow-up for any reason
* Any contraindication to CPAP use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Functional disability | 3 months
  Measured by the modified Rankin Scale, ranging from 0 (no symptoms) to 6 (death), with higher scores indicating greater disability and dependence on daily activities.

SECONDARY OUTCOMES:
Neurological impairment | Admission, 72 hours, day 5/discharge, 3 months, and 6 months
  Stroke severity will be measured by National Institutes of Health Stroke Scale, which ranges from 0 to 42, with higher scores reflecting greater neurological impairment. Neurological deterioration was defined as an increase of 4 or more points on the NIH Stroke Scale within 72 hours after stroke onset
Functional independence | Day 5/discharge, 3 months, 6 months, 1 year, and 2 years
  Measured by the modified Rankin Scale (dichotomized analysis with mRS ≤ 2) and the Barthel Index, which ranges from 0 (worst, fully dependent) to 100 (best, independent).
Cognitive impairment | Day 5/discharge, 3 months, 1 year, and 2 years
  Evaluated through the Montreal Cognitive Assessment, which was developed as a brief screening instrument for mild cognitive impairment. It assesses different cognitive domains, scoring up to 30.
Subjective quality of life | Day 5/discharge, 3 months, 6 months, 1 year, and 2 years
  Measured by the EuroQol-5 Dimension (no problems = 1; some problems = 2; and extreme problems or unable to = 3).
Depressive episode | Day 5/discharge, 3 months, 1 year, and 2 years
  Assessed using the MINI-International Neuropsychiatric Interview, which is a structured interview to assess symptoms related to depression. Questions are phrased to allow only "yes" or "no" answers.
Excessive daytime sleepiness | Admission, 3 months, 6 months, 1 year, and 2 years
  Assessed using the Epworth Sleepiness Scale. The total score, calculated by adding up the values of each answer, ranges from 0 to 24. A score of 10 or higher indicates excessive daytime sleepiness.
Mortality | 2 years
  Mortality resulting from any cause will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas, Ribeirão Preto Medical School, University of São Paulo, Ribeirão Preto, São Paulo, Brazil